CLINICAL TRIAL: NCT04288102
Title: A Phase II, Multicenter, Randomized, Double-blind, Placebo-controlled Trial to Evaluate the Efficacy and Safety of Human Umbilical Cord-derived Mesenchymal Stem Cells in the Treatment of Severe COVID-19 Patients
Brief Title: Treatment With Human Umbilical Cord-derived Mesenchymal Stem Cells for Severe Corona Virus Disease 2019 (COVID-19)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Beijing 302 Hospital (Other)
Collaborators: Huoshenshan Hospital (Other); Maternal and Child Health Hospital of Hubei Province (Other); The General Hospital of Central Theater Command (Other); Vcanbio Cell and Gene Engineering Corp., Ltd. (Industry)
Responsible Party: Principal Investigator, Fu-Sheng Wang, Head of Treatment and Research Center for Infectious Diseases, Principle Investigator, Clinical Professor, Beijing 302 Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2020-013-D
Record Dates: First submitted 2020-02-24; First posted 2020-02-28 (Actual); Last update posted 2020-08-19 (Actual); Status verified 2020-08

CONDITIONS: Corona Virus Disease 2019(COVID-19)

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, placebo-controlled study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Human Umbilical Cord-Mesenchymal Stem Cells (UC-MSCs) (Experimental): Participants will receive standard of care plus 3 does of UC-MSCs
  Interventions: Biological: UC-MSCs
- Placebo (Placebo Comparator): Participants will receive standard of care plus 3 does of placebo
  Interventions: Biological: Saline containing 1% Human serum albumin（solution without UC-MSCs）

INTERVENTIONS:
Biological: UC-MSCs — 3 does of UC-MSCs(4.0*10E7 cells per time) intravenously at Day 0, Day 3, Day 6.
  Arms: Human Umbilical Cord-Mesenchymal Stem Cells (UC-MSCs)
Biological: Saline containing 1% Human serum albumin（solution without UC-MSCs） — 3 does of placebo（intravenously at Day 0, Day 3, Day 6）
  Arms: Placebo

SUMMARY:
COVID-19 caused clusters of severe respiratory illness and was associated with 2% mortality. No specific anti-viral treatment exists. The mainstay of clinical management is largely symptomatic treatment, with organ support in intensive care for seriously ill patients. Cellular therapy, using mesenchymal stem cells has been shown to reduce nonproductive inflammation and affect tissue regeneration and is being evaluated in patients with ARDS. This clinical trial is to inspect the safety and efficiency of mesenchymal stem cells (MSCs) therapy for severe COVID-19.

DETAILED DESCRIPTION:
The Corona Virus Disease 2019 (COVID-19) caused by severe acute respiratory syndrome corona virus 2 (SARS-CoV-2) infection has unprecedentedly spread in the worldwide and been declared as a pandemic by the world health organization. COVID-19 is characterized by sustained cytokines production and hyper-inflammation, can cause clusters of severe respiratory illness with a fatality rate around 2-5%. There are currently no prophylactic vaccine and no specific antiviral treatment agents available recommended for COVID-19. Therefore, it is urgent to find a safe and effective therapeutic approach to COVID-19.

During the last decade, the promising features of mesenchymal stem cells (MSCs), including their regenerative properties and ability to differentiate into diverse cell lineages, have generated great interest among researchers whose work has offered intriguing perspectives on cell-based therapies for various diseases. These findings seem to highlight that the beneficial effect of MSC-based treatment could be principally due by the immunomodulation and regenerative potential of these cells. MSCs could significantly reduce the pathological changes of lung and inhibit the cell-mediated immune inflammatory response induced by influenza virus in animal model . MSCs has been shown to reduce nonproductive inflammation and affect tissue regeneration and is being evaluated in patients with ARDS. Our phase I preliminary data of parallel assignment study(NCT04252118) showed that three doses of MSCs was safe in patients with COVID-19. Randomized control trial is needed to assess efficacy and safety.

The investigators will do a prospective, double-blind, multicentre, randomised trial to assess treatment with three intravenous doses of MSCs compared with placebo. 90 severe COVID-19 patients will be recruited in China. 60 patients will receive i.v. transfusion 3 times of MSCs (4.0*10E7 cells per time) and the standard of care as the treated group. In addition, the 30 patients will receive placebo and standard of care as control group.

Change in lesion proportion (%) of full lung volume from baseline to day 10, day28 and 90, change in consolidation/ ground-glass lesion proportion (%) of full lung volume from baseline to day 10, 28 and 90, time to clinical improvement in 28 days, mMRC (Modified Medical Research Council) dyspnea scale, 6-minute walk test, maximum vital capacity (VCmax), Diffusing Capacity (DLCO), oxygen saturation, oxygenation index, duration of oxygen therapy, side effects, immunological characteristics (immune cells, inflammatory factors, etc.) will be evaluated during the 90 days follow up.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, aged at 18 years (including) -75 years old
2. Hospitalized
3. Laboratory confirmation of SARS-CoV-2 infection by reverse-transcription polymerase chain reaction (RT-PCR) from any diagnostic sampling source
4. Pneumonia that is judged by computed tomography
5. In accordance with any one of the following : 1)dyspnea (RR ≥ 30 times / min), 2)finger oxygen saturation ≤ 93% in resting state, 3)arterial oxygen partial pressure (PaO2) / oxygen absorption concentration (FiO2) ≤ 300MMHG, 4)pulmonary imaging shows that the focus progress > 50% in 24-48 hours
6. Interstitial lung damage is judged by computed tomography.

Exclusion Criteria:

1. Pregnancy, lactation and those who are not pregnant but do not take effective contraceptives measures;
2. Patients with malignant tumor, other serious systemic diseases and psychosis;
3. Patients who are participating in other clinical trials;
4. Inability to provide informed consent or to comply with test requirements.
5. Co-Infection of HIV, tuberculosis, influenza virus, adenovirus and other respiratory infection virus.
6. Invasive ventilation
7. Shock
8. Combined with other organ failure( need organ support)
9. Interstitial lung damage caused by other reasons ( in 2 weeks)
10. The pulmonary imaging revealed the interstitial damage of lungs before the COVID-19 confirmed.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2020-03-05 (Actual); Primary Completion 2020-05-12 (Actual); Study Completion 2020-07-09 (Actual)

PRIMARY OUTCOMES:
Change in lesion proportion (%) of full lung volume from baseline to day 28. | Day 28
  Evaluation of Pneumonia Improvement

SECONDARY OUTCOMES:
Change in lesion proportion (%) of full lung volume from baseline to day 10 and 90 | Day 10, Day 90
  Evaluation of Pneumonia Improvement
Change in consolidation lesion proportion (%) of full lung volume from baseline to day 10, 28 and 90. | Day 10, Day 28, Day 90
  Evaluation of Pneumonia Improvement
Change in ground-glass lesion proportion (%) of full lung volume from baseline to day 10, 28 and 90. | Day 10, Day 28, Day 90
  Evaluation of Pneumonia Improvement
Pulmonary fibrosis - related morphological features in CT scan at day 90 a. cord-like shadow b. honeycomb-like shadows c. interlobular septal thickening d. intralobular interstitial thickening e. pleural thickening | Day 90
  Evaluation of Pneumonia Improvement
Lung densitometry: Change in total voxel 'weight' in lesion area voxel 'weight'=voxel density (in HU) × voxel volume (in voxel) | Day 10, Day 28, Day 90
  Evaluation of Pneumonia Improvement
Lung densitometry: volumes histogram of lung density distribution (<-750, -750~-300, -300~50, >50) at day 10, 28 and 90. | Day 10, Day 28, Day 90
  Evaluation of Pneumonia Improvement
Time to clinical improvement in 28 days. | Day 28
  Clinical improvement defined as a one-point deduction from baseline in a 6 ordinal scale:
  1. Not hospitalized;
  2. Hospitalized, not requiring supplemental oxygen;
  3. Hospitalized, requiring supplemental oxygen;
  4. Hospitalized, on non-invasive ventilation or high flow oxygen devices;
  5. Hospitalized, on invasive mechanical ventilation or ECMO;
  6. Death.
Oxygenation index( PaO2/FiO2) | Day 6, Day 10, Day 28
  Evaluation of Pneumonia Improvement
Duration of oxygen therapy(days) | Day 28, Day 90
  Evaluation of Pneumonia Improvement
Blood oxygen saturation | Day 6, Day 10, Day 28
  Evaluation of Pneumonia Improvement
6-minute walk test | Day 28, Day 90
  Evaluation of Pneumonia Improvement
Maximum vital capacity (VCmax) | Baseline, Day 10, Day 14, Day 21, Day 28, Day 90
  Evaluation of Pneumonia Improvement
Diffusing Capacity (DLCO) | Baseline, Day 10, Day 14, Day 21, Day 28, Day 90
  Evaluation of Pneumonia Improvement
mMRC (Modified Medical Research Council) dyspnea scale | Day 28, Day 90
  Evaluation of Pneumonia Improvement
  No limitation of activities, discharged from hospital =Score 1; Hospitalized, no oxygen therapy=Score 2; Oxygen by mask or nasal prongs-Score 3; Non-invasive ventilation or high-flow oxygen=Score 4; Mechanical ventilation or ECMO=Score 5; Death=Score 6.
Changes of absolute lymphocyte counts and subsets from baseline to day 6, 10, 28 and 90. | Day 6, Day 10, Day 28, Day 90
  Marker of Immunological function
Changes of cytokine/chemokine levels from baseline to day 6, 10, 28 and 90. | Day 6, Day 10, Day 28, Day 90
  Marker of Immunological function
Adverse events | Day 0 through Day 90
  Safety endpoints
Serious adverse events | Day 0 through Day 90
  Safety endpoints
All-cause mortality | Day 0 through Day 90
  Safety endpoints

CONTACTS AND LOCATIONS:
Overall Officials: Fu-Sheng Wang, MD, PhD, Study Chair — Beijing 302 Hospital
Locations (3):
- China (3):
  - General Hospital of Central Theater Command, Wuhan, Hubei
  - Maternal and Child Hospital of Hubei Province, Wuhan, Hubei
  - Wuhan Huoshenshan Hospital, Wuhan, Hubei

IPD SHARING:
Plan to Share IPD: Yes
After approval from the steering committee and the Human Genetic Resources Administration of China, this trial data can be shared with qualifying researchers who submit a proposal with a valuable research question. A contract should be signed.

REFERENCES:
- [Derived] Yuan MQ, Song L, Wang ZR, Zhang ZY, Shi M, He J, Mo Q, Zheng N, Yao WQ, Zhang Y, Dong T, Li Y, Zhang C, Song J, Huang L, Xu Z, Yuan X, Fu JL, Zhen C, Cai J, Dong J, Zhang J, Xie WF, Li Y, Zhang B, Shi L, Wang FS. Long-term outcomes of mesenchymal stem cell therapy in severe COVID-19 patients: 3-year follow-up of a randomized, double-blind, placebo-controlled trial. Stem Cell Res Ther. 2025 Feb 25;16(1):94. doi: 10.1186/s13287-025-04148-1. PMID 40001244
- [Derived] Li TT, Zhang B, Fang H, Shi M, Yao WQ, Li Y, Zhang C, Song J, Huang L, Xu Z, Yuan X, Fu JL, Zhen C, Zhang Y, Wang ZR, Zhang ZY, Yuan MQ, Dong T, Bai R, Zhao L, Cai J, Dong J, Zhang J, Xie WF, Li Y, Shi L, Wang FS. Human mesenchymal stem cell therapy in severe COVID-19 patients: 2-year follow-up results of a randomized, double-blind, placebo-controlled trial. EBioMedicine. 2023 Jun;92:104600. doi: 10.1016/j.ebiom.2023.104600. Epub 2023 May 5. PMID 37149930
- [Derived] Shi L, Yuan X, Yao W, Wang S, Zhang C, Zhang B, Song J, Huang L, Xu Z, Fu JL, Li Y, Xu R, Li TT, Dong J, Cai J, Li G, Xie Y, Shi M, Li Y, Zhang Y, Xie WF, Wang FS. Human mesenchymal stem cells treatment for severe COVID-19: 1-year follow-up results of a randomized, double-blind, placebo-controlled trial. EBioMedicine. 2022 Jan;75:103789. doi: 10.1016/j.ebiom.2021.103789. Epub 2021 Dec 25. PMID 34963099
- [Derived] Shi L, Huang H, Lu X, Yan X, Jiang X, Xu R, Wang S, Zhang C, Yuan X, Xu Z, Huang L, Fu JL, Li Y, Zhang Y, Yao WQ, Liu T, Song J, Sun L, Yang F, Zhang X, Zhang B, Shi M, Meng F, Song Y, Yu Y, Wen J, Li Q, Mao Q, Maeurer M, Zumla A, Yao C, Xie WF, Wang FS. Effect of human umbilical cord-derived mesenchymal stem cells on lung damage in severe COVID-19 patients: a randomized, double-blind, placebo-controlled phase 2 trial. Signal Transduct Target Ther. 2021 Feb 10;6(1):58. doi: 10.1038/s41392-021-00488-5. PMID 33568628